CLINICAL TRIAL: NCT03995719
Title: Study to Assess the Impact of an Educational Program for Ostomy Patients (Ostomeducat)
Brief Title: Educational Program for Ostomy Patients (Ostomeducat)
Acronym: ostomeducat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mª Victoria Maestre Sanchez (Other)
Collaborators: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Sponsor-Investigator, Mª Victoria Maestre Sanchez, Sponsor-Investigator, Hospitales Universitarios Virgen del Rocío
Organization: Hospitales Universitarios Virgen del Rocío (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EPOP2018
Record Dates: First submitted 2019-04-30; First posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Educational Problems; Colostomy Complications; Surgery; Colorectal Disorders
Keywords: colostomy; education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative education (Other): Each patient had individual consultation several days before surgery with the stoma nurse specialist, following standard ostomy teaching plans
  Interventions: Other: Preoperative education; Other: Postoperative education
- Postoperative education (Other): Each patient had individual consultationseveral days before surgery with the stoma nurse specialist, following standard ostomy teaching plans
  Interventions: Other: Preoperative education; Other: Postoperative education

INTERVENTIONS:
Other: Preoperative education — 65 patients were instructed to a preoperative stoma-education program
Other: Postoperative education — 73 patients, receiving the same information in postoperative period.

SUMMARY:
Stoma surgery is a relatively common treatment for patients suffering from colorectal diseases.This study aimed to investigate the impact on hospital stay and short-term overall complications prior to and following the introduction of an outpatient preoperative stoma education program.

DETAILED DESCRIPTION:
38 patients undergoing stoma surgery were analyzed, 73 prior education program and 65 following it.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age undergoing elective colorectal resections that eventually would require formation of a stoma (colorectal cancer up to 20 cm from the anal verge, colonic poliposis and inflammatory bowel disease).

Exclusion Criteria:

* Patients already had a stoma before the operation or in case of emergent surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of.complications | First 30 days after surgery
  Surgical complications
Rate of mortality (assessed by Clavien-Dindo Classification) | First 30 days after surgery
  Patient mortality within the first 30 days after surgery

SECONDARY OUTCOMES:
Rate of readmissions | the first 30 days after surgery
  Number of patient hospitalization within the first 30 days after surgery
Reinterventions | 30 days after surgery
  Patient new surgery

CONTACTS AND LOCATIONS:
Overall Officials: ANA Mª GARCIA CABRERA, PHD, Principal Investigator — coloproctology unit
Locations (1):
- Hospital Universitario Virgen Del Rocio, Seville, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
Publishing
Supporting Information: Study Protocol
Time Frame: between July 2014 and June 2015
Access Criteria: patients older than 18 years of age undergoing elective colorectal resections that eventually would require formation of a stoma (colorectal cancer up to 20 cm from the anal verge, colonic poliposis and inflammatory bowel disease).
  Patients were excluded from the study if they already had a stoma before the operation or in case of emergent surgery.

REFERENCES:
- [Derived] Garcia-Cabrera AM, de la Portilla de Juan F, Navarro-Morales L, Ribera Garcia S, Duran Ventura MDC, Fernandez Luque I, Padillo-Ruiz FJ. Influence of Preoperative Educational Intervention for Patients Undergoing Fecal Ostomy Surgery: A Comparison Cohort Study. J Wound Ostomy Continence Nurs. 2023 Nov-Dec 01;50(6):484-488. doi: 10.1097/WON.0000000000001020. PMID 37966076

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT03995719/Prot_SAP_000.pdf